CLINICAL TRIAL: NCT01609374
Title: Prospective, Non-Randomized, Concurrently Controlled, Multi-Center Study to Evaluate the Safety and Effectiveness of the Spinal Kinetics™ M6-C Artificial Cervical Disc Compared to Anterior Cervical Discectomy and Fusion (ACDF) for the Treatment of Symptomatic Cervical Radiculopathy
Brief Title: Restore CLINICAL TRIAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Spinal Kinetics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-C002
Record Dates: First submitted 2012-05-24; First posted 2012-06-01 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-03

CONDITIONS: Cervical Radiculopathy; Degenerative Disc Disease
Keywords: Spinal Kinetics; artificial cervical disc; cervical radiculopathy; ACDF; neck pain; cervical spine; degenerative disc disease
MeSH Terms: conditions — Radiculopathy; Intervertebral Disc Degeneration; Neck Pain

STUDY DESIGN:
Intervention Model Description: non-randomized, concurrent ACDF control
Masking Description: since the study is concurrently controlled, masking is not possible
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- M6-C Artificial Cervical Disc (Experimental)
  Interventions: Device: M6-C Artificial Cervical Disc
- Anterior Cervical Discectomy and Fusion (Active Comparator)
  Interventions: Device: Anterior plate system with corticocancellous allograft bone

INTERVENTIONS:
Device: M6-C Artificial Cervical Disc — Total disc replacement
  Arms: M6-C Artificial Cervical Disc
Device: Anterior plate system with corticocancellous allograft bone — Cervical fusion
  Arms: Anterior Cervical Discectomy and Fusion

SUMMARY:
This is a prospective, concurrently controlled, multi-center study to evaluate the safety and effectiveness of the Spinal Kinetics M6-C artificial cervical disc compared to anterior cervical discectomy and fusion (ACDF) for the treatment of symptomatic cervical radiculopathy with or without cord compression. Some participating sites will enroll just M6-C patients, while others will enroll just ACDF patients.

Patients eligible for study enrollment will present with degenerative cervical radiculopathy requiring surgical intervention, confirmed clinically and radiographically, at one vertebral level from C3 to C7.

A total of 243 subjects will be included at up to 20 sites.

ELIGIBILITY:
All study subjects must present with degenerative cervical radiculopathy with or without spinal cord compression, confirmed clinically and radiologically, requiring surgical intervention at a single vertebral level from C3 to C7.

Inclusion Criteria:

1. Diagnosis of degenerative cervical radiculopathy with or without spinal cord compression requiring surgical treatment at one level from C3 to C7 demonstrated by signs and/or symptoms of disc herniation and/or osteophyte formation (e.g. neck and/or arm pain, radiculopathy, etc.) and is confirmed by patient history and radiographic studies (e.g. MRI, CT, x-rays, etc.)
2. Inadequate response to conservative medical care over a period of at least 6 weeks
3. Neck Disability Index score of ≥ 30% (raw score of ≥ 15/50)
4. Neck or arm pain VAS ≥ 4 on a scale of 0 to 10
5. Willing and able to comply with the requirements of the protocol including follow-up requirements
6. Willing and able to sign a study specific informed consent
7. Skeletally mature and ≥ 18 years old and ≤ 75 years old

Exclusion Criteria:

1. More than one cervical level requiring surgery
2. Previous anterior cervical spine surgery
3. Axial neck pain as the solitary symptom
4. Previous posterior cervical spine surgery (e.g., posterior element decompression) that destabilizes the cervical spine
5. Advanced cervical anatomical deformity (e.g., ankylosing spondylitis, scoliosis) at the operative or adjacent levels
6. Symptomatic facet arthrosis
7. Less than 4º of motion in flexion/extension at the index level
8. Instability as evidenced by subluxation > 3 mm at the index or adjacent levels as indicated on flexion/extension x-rays
9. Advanced degenerative changes (e.g., spondylosis) at the index vertebral level as evidenced by bridging osteophytes, central disc height < 4mm and/or < 50% of the adjacent normal intervertebral disc, or kyphotic deformity > 11º on neutral x-rays
10. Severe cervical myelopathy (i.e., Nurick's Classification > 2)
11. Active systemic infection or infection at the operative site
12. Co-morbid medical conditions of the spine or upper extremities that may affect the cervical spine neurological and/or pain assessment
13. Metabolic bone disease such as osteoporosis that contradicts spinal surgery (for females over 50 and males over 55 years old, or if the score on the Osteoporosis Self-Assessment Test is < 2, a dual energy x-ray absorptiometry [DEXA scan] of the spine is required; if the bone mineral density T-score in the spine is ≤ -2.5 the patient must be excluded)
14. History of an osteoporotic fracture of the spine, hip or wrist
15. History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism
16. Taking medications that may interfere with bony/soft tissue healing including chronic steroid use
17. Known allergy to titanium, stainless steels, polyurethane, polyethylene, or ethylene oxide residuals
18. Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C or fibromyalgia
19. Insulin-dependent type 1 or type 2 diabetes
20. Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion
21. Pregnant, or intend to become pregnant, during the course of the study
22. Severe obesity (Body Mass Index > 40)
23. Physical or mental condition (e.g., psychiatric disorder, senile dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain or quality of life.
24. Involved in current or pending spinal litigation where permanent disability benefits are being sought
25. Incarcerated at the time of study enrollment
26. Current participation in other investigational study that may impact study outcomes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation through 24 months | 24 months
  Evaluate the safety by assessing adverse events and neurological function following implantation with the Spinal Kinetics M6-C artificial cervical disc compared to anterior cervical discectomy and fusion (ACDF)
Effectiveness Evaluation through 24 months | 24 months
  Evaluate the effectiveness using Neck Disability Index (NDI)

SECONDARY OUTCOMES:
Effectiveness of the Spinal Kinetics M6-C artificial cervical disc compared to anterior cervical discectomy and fusion (ACDF) | 6 weeks, 3 months, 6 months, 12 months, 24 months
  Evaluate the Neck and Arm pain VAS, health-related quality of life SF-36, surgery outcomes, patient satisfaction and quantitative and qualitative radiographic assessments